CLINICAL TRIAL: NCT04864067
Title: No Operation After Short Course Equivalent Dose (Ht) Radiation Therapy Followed By Consolidation Chemotherapy In Locally Advanced Rectal Cancer: The Prospective, Single Arm NOAHS-ARC Trial
Brief Title: No Operation After Short Course Radiotherapy Followed By Consolidation Chemotherapy In Locally Advanced Rectal Cancer
Acronym: NOAHS-ARC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Servicio de Salud Metropolitano Sur Oriente (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FONDECYT 11201291
Record Dates: First submitted 2021-04-25; First posted 2021-04-28 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Radiotherapy; Neoadjuvant therapy; Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms; Adenocarcinoma | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Capecitabine; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Short Course Radiotherapy and Consolidation Chemotherapy (Experimental): This arm will receive short course radiotherapy (5x5 Gy) during 1 week. Between 7 to 14 days after radiotherapy, patient will receive 9 cycles of FOLFOX. CapeOX may be given as alternative for FOLFOX.
  Interventions: Drug: Oxaliplatin; Drug: 5-Fluoracil; Drug: Leucovorin; Drug: Capecitabine; Radiation: 5x5 Gy; Behavioral: Quality of Life Questionnaires; Procedure: DRE/ Endoscopy

INTERVENTIONS:
Drug: Oxaliplatin — Consolidation Chemotherapy
  Other Names: All Brands
Drug: 5-Fluoracil — Consolidation Chemotherapy
  Other Names: All Brands
Drug: Leucovorin — Consolidation Chemotherapy
  Other Names: All Brands
Drug: Capecitabine — Consolidation Chemotherapy
  Other Names: All Brands
Radiation: 5x5 Gy — Neoadjuvant Radiotherapy
Behavioral: Quality of Life Questionnaires — Quality of Life Evaluation (LARS Score, IIEF, FSFI, I-PSS and EORTC QLQ-C30)
Procedure: DRE/ Endoscopy — Flexible Sigmoidoscopy and Digital Rectal Exam

SUMMARY:
This study is designed to explore the hypothesis that in patients with a Locally advanced rectal cancer (LARC) treated with a Total neoadjuvant therapy (TNT) strategy based on short course radiotherapy (5x5Gy) followed by neoadjuvant consolidation chemotherapy is associated with a higher rate of pathological clinical response and sustained (>1year) complete clinical response when compared to an historical cohort treated with long course chemoradiation therapy (CRT), total mesorectal excision (TME) and adjuvant chemotherapy (ACT).

DETAILED DESCRIPTION:
Non-operative management with a Watch and Wait (W&W) strategy has been advocated for selected patients with a locally advanced rectal cancer (LARC) and a complete clinical response (cCR) after neoajuvant (NA) treatment.

In this context, total neoadjuvant therapy (TNT), i.e the use of radiotherapy and full dose of post-operative chemotherapy as part of NA treatment, has emerged as a strategy to enhance treatment response.

Currently, TNT has reported higher rates of pCR and organ preservation when compared to current standard of care. However, the best TNT strategy is still unknown. We therefore hypothesize that in LARC patients, the use of a TNT strategy based on short course RT followed by consolidation chemotherapy is associated with a higher rate of pCR and sustained (>1year) cCR when compared to an historic cohort.

The main aim of the present proposal is to assess the effects of a standardized TNT model in LARC patients as a strategy for enhanced pCR/sustained cCR. For this purpose, we propose the following experimental model: In primary Aim 1 we will study if the effects of a TNT strategy over patients with a LARC enhance the rate of pCR/sustained cCR by (1) evaluating the compliance and toxicity of a TNT strategy as a proof of concept of its applicability, (2) assessing the rate of cCR at the end of TNT and (3) assessing the rate of pCR in the surgically managed subgroup and sustained cCR (>1year) in the W&W subgroup. Additionally, in primary Aim 2, we will determine if patients with a W&W strategy have better functional outcomes and quality of life (QoL) than patients treated with TME after TNT by (1) using validated questionnaires for the evaluation of bowel, sexual and urinary function for W&W and TME patients and (2) by evaluating the QoL using a widely-used standardized questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the rectum
* Clinical Stage II (T3-4, N-) or Stage III (any T, N+) based on Magnetic Resonance Imaging (MRI)
* Tumors < 7cm from anal verge (palpable)
* No prior history of rectal cancer

Exclusion Criteria

* Patients with tumors >7cm from anal verge
* ECOG >1,
* Contraindication for chemotherapy: Hemoglobin <8, White Blood Count <4000, Platelets <100,000, Creatinine Clearance <50ml/min, Total Bilirubin <5mg/dl,
* Stage IV at diagnosis
* Coronary artery disease, either no treated or recent acute coronary syndrome in the last 12 months.
* Congestive heart failure
* Peripheral neuropathy
* Previous pelvic radiotherapy
* Prior rectal cancer treatment
* Pregnancy or nursery
* Any contraindications to MRI (e.g. patients with pacemakers)
* Indication of pelvic exenteration
* Impossibility to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of pathological and sustained clinical response | 3 years
  Combined number of patients with pathological response in the surgical specimen and patients in a Watch and Wait protocol with a sustained clinical response longer than a year.
Quality of Life and Funcional Outcomes | 3 years
  Standardized evaluation using validated questionnaires comparing patients undergoing TME versus WW patients in the cohort

SECONDARY OUTCOMES:
Adverse events | 3 years
  Adverse events will be graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe F Quezada-Diaz, MD, Principal Investigator — Complejo Asistencial Doctor Sótero del Rio; Nicole M Caire, MD, Principal Investigator — Complejo Asistencial Doctor Sótero Del Río
Locations (3):
- Chile (3):
  - Complejo Asistencial Doctor Sótero del Rio, Santiago, RM
  - Hospital La Florida, Santiago, RM
  - Hospital Padre Hurtado, Santiago, RM

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quezada-Diaz FF, Bercz A, Escobar JL, Caire N, Diaz-Feldman LE, Manriquez E, Carvajal G. No operation after short-course radiotherapy followed by consolidation chemotherapy in locally advanced rectal cancer (NOAHS-ARC): study protocol for a prospective, phase II trial. Int J Colorectal Dis. 2025 Mar 18;40(1):69. doi: 10.1007/s00384-025-04850-9. PMID 40100473